CLINICAL TRIAL: NCT02687880
Title: Testicular Tissue Cryopreservation for Fertility Preservation in Male Patients Facing Infertility-causing Diseases or Treatment Regimens
Status: Withdrawn | Type: Observational
Why Stopped: Prior to start up, study was discontinued for feasibility reasons
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-2047
Record Dates: First submitted 2016-02-18; First posted 2016-02-22 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Infertility; Cryopreservation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will provide a pool of research tissue that will be used to develop and test methods for manipulation and cryopreservation of testicular tissue. Progress in these investigations may open up a range of new fertility preservation techniques to patients that currently have no options. At the same time, a substantial portion of the patient's tissue will be cryopreserved and reserved for his own future use.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Subjects: All subjects will undergo a surgical procedure (Testicular biopsy) to harvest their testicular tissue. In most cases, this will be done as part of their routine care but it is possible the subject may elect to have the procedure as part of a "research only" biopsy.
  Interventions: Procedure: Testicular biopsy

INTERVENTIONS:
Procedure: Testicular biopsy — Subjects will undergo a surgical procedure to harvest their testicular tissue.

SUMMARY:
Many chemotherapy and radiation-containing regimens for cancer or prior to bone marrow transplantation can cause sterility in children and young adults. In addition, some human disease conditions (e.g., Klinefelter's) are associated with infertility. Semen cryopreservation is available as a fertility-preserving option for post pubertal boys and adult men, but many do not take advantage of this option due in part to lack of information, illness, and/or time constraints relative to their treatment plan. Currently, no fertility-preserving options are available for prepubescent boys who are not yet producing sperm. The primary objective of the proposed study is to 1) Optimize techniques for cryopreserving testicular tissue, 2) Assess malignant contamination in testicular tissues and 3) develop methods to enrich spermatogonial stem cells and remove malignant contamination from testicular tissue. In addition, this study will process and cryopreserve tissue and/or cells for participating patients as a resource for future elective procedures to attempt fertility restoration.

ELIGIBILITY:
Inclusion Criteria:

1. Male age 30 days (non-inclusive) to 39 years (inclusive).
2. Scheduled to undergo surgery, chemotherapy, drug treatment and/or radiation for the treatment or prevention of a medical condition or malignancy with risk of causing permanent and complete loss of subsequent testicular function.
3. Have a medical condition or malignancy that requires removal of all or part of one or both testicles.
4. Have newly diagnosed or recurrent disease.

   a) Those who were not enrolled at the time of initial diagnosis (i.e., patients with recurrent disease) are eligible if they have not previously received therapy that is viewed as likely to result in complete and permanent loss of testicular function.
5. Have two testicles if undergoing elective removal of a testicle for fertility preservation only.

   b) Note: removal of both testicles will limit fertility preservation options.
6. Fully executed approved informed consent and authorization permitting the release of personal health information.

   c) The patient and/or the patient's legally authorized guardian must acknowledge in writing that consent for specimen collection has been obtained, in accordance with institutional policies approved by the U.S. Department of Health and Human Services.
7. Consent for serum screening tests for infectious diseases [HIV-1, HIV-2, hepatitis B, hepatitis C, RDR (syphilis), CMV, HLTV-1, and HTLV-2], to be performed at the time of testicular tissue harvesting.
8. Undergo a full history and physical examination.
9. Obtain standard pre-operative clearance (based on the most recent ACC/AHA Guideline for Perioperative Cardiovascular Evaluation for Noncardiac Surgery) as determined by their primary surgeon.

Exclusion Criteria:

1. Diagnosed with psychological, psychiatric, or other conditions which prevent giving fully informed consent.
2. Diagnosed with an underlying medical condition that significantly increases their risk of complications from anesthesia and surgery.

Ages: 31 Days to 39 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Males scheduled to undergo surgery, chemotherapy, drug treatment and/or radiation for the treatment or prevention of a medical condition or malignancy with risk of causing permanent and complete loss of subsequent testicular function.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-12-30 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Status of frozen tissue | 1 year post-procedure
  Subjects will be contacted to determine status of frozen tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Serena Dovey, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No